CLINICAL TRIAL: NCT01884454
Title: EFFECTS OF SLEEP LOSS AND OBSTRUCTIVE SLEEP APNEA SYNDROME ON REPRODUCTIVE FUNCTION IN MEN
Brief Title: SLEEP AND OSA ON REPRODUCTIVE FUNCTION IN MEN
Acronym: PSAR01
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Monica Levy Andersen, Professor, Federal University of São Paulo
Other Study IDs: PSAR01
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep; obstructive sleep apnea; reproduction; sperm; hormones; men
MeSH Terms: conditions — Sleep Apnea, Obstructive; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Total sleep deprivation: Healthy volunteers will be submitted to total sleep deprivation (TSD) for 48 hours.
  Interventions: Behavioral: Sleep deprivation
- moderate to severe OSA: Patients diagnosed with moderate to severe obstructive sleep apnea syndrome (OSA) with normal or overweight body mass index (BMI), will be recruited.
- REM sleep deprivation: Healthy volunteers will be submitted to selective REM sleep deprivation (REMSD) for 48 hours.
  Interventions: Behavioral: Sleep deprivation
- Control: The control group will be subjects with an apnea hypopnea index <5/h.

INTERVENTIONS:
Behavioral: Sleep deprivation — Volunteers will be submitted to total sleep deprivation (SD) or selective REM sleep deprivation for 48 hours. After SD, these volunteers will be allowed to sleep for 48 hours (period rebound).
  Other Names: Total sleep deprivation; REM sleep deprivation
  Groups: REM sleep deprivation; Total sleep deprivation

SUMMARY:
In view of the hormonal changes induced by both sleep deprivation and obstructive sleep apnea syndrome (OSA), and the importance of maintaining these hormones in reproductive processes. The present study aims to evaluate the effects of the OSA or sleep deprivation (total or selective REM sleep for 48h) on reproductive function in adult men with normal body mass index.

DETAILED DESCRIPTION:
In this study will be recruited volunteers 25-50 years of age with a body mass index (BMI) 20-25 kg/m2 (normal) that after performing polysomnography, will be distributed in the following groups: healthy or diagnosed with obstructive sleep apnea syndrome (OSA). Volunteers without OSA will be submitted to total sleep deprivation (SD) or selective REM sleep deprivation for 48 hours. After SD, these volunteers will be allowed to sleep for 48 hours (period rebound). Blood samples will be taken for hormonal analysis (testosterone, luteinizing hormone, follicle-stimulating hormone, progesterone and cortisol)and gene expression. The semen collection for evaluation of sperm count (concentration, viability and sperm morphology) in three different periods, baseline collection, after SD protocols and the end of rebound period. Individuals diagnosed with OSA also have three collections of blood and semen samples for analyzes.

ELIGIBILITY:
Inclusion Criteria:

* men
* There is no discrimination of economic class
* Age between 25 and 50
* BMI 30 kg/m2
* No prior neurological, psychiatric or use of psychotropic medication
* OSA (moderate and severe apnea hypopnea index > 15)

Exclusion Criteria:

* smokers
* addiction
* Individuals with another sleep disorder
* Severe uncontrolled organic disease that might interfere with the conduct of the study, such as cancer, heart disease, digestive disorders, diabetes mellitus, male reproductive system
* Presence of moderate or severe depression and psychiatric disorders
* Volunteers with previous treatment for OSA

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  * men
  * There is no discrimination of economic class
  * Age between 25 and 50
  * BMI 30 kg/m2
  * No prior neurological, psychiatric or use of psychotropic medication
  * OSA (moderate and severe apnea hypopnea index > 15)
  Exclusion Criteria:
  * smokers
  * addiction
  * Individuals with another sleep disorder
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in sperm analysis | change from baseline, sleep deprivations and rebound period. Participants will be followed for the duration of laboratory stay, an expected average of 7 days
  - Semen collection (concentration, viability and sperm morphology)

SECONDARY OUTCOMES:
change hormonal evaluation | change from baseline, sleep deprivations and rebound period. Participants will be followed for the duration of laboratory stay, an expected average of 7 days
  - Hormonal analysis (testosterone, luteinizing hormone, follicle-stimulating hormone, progesterone and cortisol)

OTHER OUTCOMES:
Sleep patterns of the study population | Change from baseline, sleep deprivations and rebound period. Participants will be followed for the duration of laboratory stay, an expected average of 7 days
  - Polysomnography
Change gene expression | Change from baseline, sleep deprivations and rebound period. Participants will be followed for the duration of laboratory stay, an expected average of 7 days
  Blood will be collected in specific tubes (PaxGene)for RNA extraction and gene expression determination.

CONTACTS AND LOCATIONS:
Overall Officials: Tathiana A Alvarenga, PhD, Principal Investigator — Federal University of São Paulo; Monica L Andersen, Prof, Study Director — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: American Academy of Sleep Medicine — http://www.aasmnet.org/